CLINICAL TRIAL: NCT05392257
Title: Efficacy and Safety of Rituximab Plus Zanubrutinib and Lenalidomide for Relapsed and Refractory Diffuse Large B Cell Lymphoma, a Multicenter, Open and Prospective Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH20220521
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Overall Survival
MeSH Terms: interventions — Rituximab; zanubrutinib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental)
  Interventions: Drug: Rituximab + zanubrutinib + lenalidomide

INTERVENTIONS:
Drug: Rituximab + zanubrutinib + lenalidomide — Rituximab at 375mg / m2, Day 0; Zanubrutinib 160mg bid continuously oral; Lenalidomide 25mg qd oral on days 1-21; 28 days as a course of treatment

SUMMARY:
This clinical trial is an investigator-initiated multicenter, open, prospective clinical study in order to explore the efficacy and safety of rituximab plus zanubrutinib and lenalidomide in relapsed and refractory diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
Subjects are patients withRelapsed and refractory Diffuse Large B cell lymphoma (DLBCL). All included patients will be treated with rituximab plus zanubrutinib and lenalidomide. In the induction stage, patients will receive 375 mg/m2 rituximab Day 1 of Cycles 1-6, twice-daily 160 mg zanubrutinib and 25 mg lenalidomide Days 1-21 of each 28-day cycle. In the maintenance treatment period, patients will receive 375 mg/m2 rituximab every 2 months, twice-daily 160 mg zanubrutinib and 10 mg lenalidomide Days 1-21 of each 28-day cycle. Imaging evaluation will take every two cycles to determine the best therapeutic effect, PD patients will exit from the clinical trial. The comprehensive therapeutic evaluating will take after 4 cycles. Peripheral blood stem cells can be collected from young patients with PR or CR. If patients' condition is suitable after 6 cycles of induction therapies, autologous hematopoietic stem cell transplantation can be chosed for patients with PR or CR and exit from the trail.Primary study endpoint is objective response rate (ORR) at the end of 6 cycles of induction therapy. Secondary study endpoints include progression-free survival time (PFS), overall survival (OS) and adverse reaction events (TEAS). After sample size calculation, we plan to enroll 72 relapsed and refractory diffuse large B cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:1．Volunteer for clinical research; fully understand the study and sign an informed consent (ICF); be willing to follow and be able to complete all study steps; 2．Histologically confirmed diffuse large B cell lymphoma (DLBCL), and CD20-positive patients; 3．Age from 18 to 80 (patients with age > 80 and status score > 2 should be assessed by the investigator to make sure whether they are suitable for this clinical trail); 4．Relapse / refractory DLBCL, relapse or refractory disease is defined as: 1) disease recurrence after complete remission (CR), 2) partial remission (PR), disease stability (SD) or disease progression (PD) after the final treatment before the study; patients who younger than 65 should be treated with at least two different chemotherapy regimens, and patients age> 65 need at least one chemotherapy regimen, or relapse after remission; 5．Patiens have measurable lesions, the standard is showed in Appendix 1; 6．ECOG score is no more than 2; 7．The expected survival period is greater than 3 months; 8．Adequate organ and bone marrow function, no severe hematopoietic dysfunction, no cardiac, lung, liver, kidney, thyroid dysfunction, or immune deficiency (no blood transfusion, granulocyte colony stimulating factor, or other medical support drugs within 7 days prior to the start of this study) : neutrophil absolute count (ANC) ≥1.0×109/L, platelet (PLT) ≥50×109/L, hemoglobin >80 g/L, aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5×ULN, total bilirubin (TBIL) ≤1.5×ULN, creatinine clearance (Ccr) ≥40ml/min (estimated by Cockcroft-Gault formula), international standardized ratio (INR) ≤1.5×ULN, prothrombin time (PT) and activated partial thrombin time (APTT) ≤1.5×ULN (unless the subject is receiving anticoagulant therapy at screening time); 9．Patiens will be enrolled only after the toxicity of the previously treated return to 《the Common Terminology Criteria for Adverse Events》 (CTCAE) V 5.0 score<1. Irreversible toxicity caused by previous antitumor treatment and is not expected to worsen than grade 2 toxicity (e. g. thrombocytopenia, anemia, neurotoxicity, hair loss and hearing loss, during the study) should be evaluated by the investigator; 10．Patiens who do not meet the criteria for ASCT or who refuse ASCT. Patiens who relapse after ASCT can be enrolled at least 100 days after the transplantation.

11．Before starting treatment, two pregnancy tests (at least one of them should be a serological pregnancy test) should be performed and the result must be negative.The first test must be conducted within 10-14 days before lenalidomide treatment, and the second test should within 24 hours before lenalidomide treatment.

12．Fertile women must agree to use reliable contraception from 4 weeks before lenalidomide treatment to at least 90 days after the last administration of zanubrutinib and lenalidomide, or 12 months after the last administration of rituximab (whichever is longer as the standard). Male patients taking the study drug may not donate sperm throughout the study.

13．Patients are not allowed to donate blood during lenalidomide treatment and within 4weeks after withdrawal, as blood may be used in pregnant female patients whose fetus will not be exposed to lenalidomide.

Exclusion Criteria:1．Special type of lymphoma: primary mediastinal (thymus) large B cell lymphoma.

2．Patients with other hematological diseases and non-lymphoma were diagnosed. 3．Other active malignancies that require concurrent treatment. 4．Major surgery is performed within 4 weeks before screening. 5．Previous anticancer therapy toxicity is still equal to or more than grade 2 when enrol (except for alopecia, ANC, hemoglobin and platelet toxicity); ANC, hemoglobin and platelet-related requirements, please follow the inclusion criteria 9.

6．History of other active malignant diseases within 2 years prior to study entry, but the following situation are eligibility for inclusion: 1) adequately treated carcinoma in situ of the cervix; 2) Local basal cell carcinoma or squamous cell carcinoma of the skin; 3) Pre-existing malignant disease that has been controlled and treated locally and radically (surgically or otherwise).

7．Have clinically significant cardiovascular disease, including: 1) myocardial infarction that occurred within 6 months prior to screening stage; 2) Unstable angina pectoris within 3 months before screening stage; 3) Clinical major arrhythmia (e.g., persistent ventricular tachycardia, ventricular fibrillation, tachycardia with torsional tip); 4) QTcF (corrected according to Fridericia formula) >480 msec; 5) History of second-degree type II atrioventricular block or third-degree ATrioventricular block; 6) Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA).

8．History of severe hemorrhagic disease, such as hemophilia A, hemophilia B, von willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.

9．History of stroke or intracranial hemorrhage within 6 months prior to the first taking of the investigational drug.

10．Inability to swallow capsules or a medical condition that significantly affects gastrointestinal function, such as malabsorption syndrome, gastrectomy or small bowel resection, symptomatic inflammatory bowel disease, or partial or complete intestinal obstruction; 11．Uncontrolled systemic infection requiring intravenous administration of drugs for parenteral anti-infective therapy.

12．Human immunodeficiency virus (HIV) infection, or presence of serological status of active hepatitis B or C virus infection: 1）Either hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive serology can be enrolled if hepatitis B virus (HBV) DNA (<20 IU/mL) and are willing to receive monthly HBV reactivation monitoring. 2) For patients in the presence of hepatitis C virus antibody, they could be enrolled if HCV RNA is not detected.

13．Hypersensitivity is known to either lenalidomide or rituximab, or to chemical or biological analogues of lenalidomide and rituximab.

14．Women during pregnancy or lactation. 15．Any life-threatening disease, medical condition, or incomplete organ system as considered by the investigator that may affect the safety of the subject or lead to the study risk.

16．History of deep venous thrombosis (DVT) or pulmonary embolism (PE) in the past 12 months.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The overall survival in this population of patients | 24 months
  The overall survival of the enrolled patients from start the combination treatment of Rituximab + zanubrutinib + lenalidomide regimen

SECONDARY OUTCOMES:
The progression free survival in this population of patients | 24 months
  The progression free survival of the enrolled patients from start the combination treatment of Rituximab + zanubrutinib + lenalidomide regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao central Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR